CLINICAL TRIAL: NCT04040283
Title: Platelet-rich Plasma for Menical Tear
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Ivan Medina-Porqueres, Professor, University of Malaga
Other Study IDs: UMalaga21
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Platelet-Rich Plasma; Meniscus Lesion
Keywords: Growth factors; Meniscal injury
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Platelet-rich plasma (PRP) therapy — Platelet rich plasma (PRP) describes a technique in which platelets are isolated from a sample of a person's own blood using simple cell-separating systems such as centrifugation in order to obtain highly concentrated samples of platelets that can be re-injected into an injury site to promote healing.

SUMMARY:
Meniscal injuries are a common pathology among athletes, and have an impact on the daily or sporting practice of patients. Surgical approach implies sometimes heavy consequences. Platelet-rich-plasma (PRP) has been shown to be effective in accelerating wound healing and tissue regeneration in orthopedic and oral surgery. This clinical trial aims to investigate the safety and efficacy of intraarticular and periferal PRP injection in patients with stable meniscal injury. The pre- and post-interventional clinical outcomes will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients 18-70 years of age
* With diagnosis of meniscus injury
* Single tear of the medial and/or lateral meniscus
* With no indication of meniscus repair surgery

Exclusion Criteria:

* Prior history of multiple ligaments injury, associated significant ligament instability: Grade III MCL, Grade III PCL, or ACL deficient knee
* Prior history of knee surgery
* Discoid meniscus
* Osteoarthritic changes (Kellgren Lawrence scale >2)
* Inflammatory diseases (i.e. rheumatoid arthritis)
* Underlying bleeding disorder or coagulopathy
* Concominant chondral defects (> 2 ICRS)
* Cancer patients
* Pregnancy
* Patients who will not cooperate with six-month followup

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Skeletally mature patients aged between 18 and 70 years with imaging and clinical diagnosis of meniscus injury and no indication of meniscus repair surgery
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score scale | 6months post procedure
Visual Analog Scale | 6months post procedure

SECONDARY OUTCOMES:
International Knee Documentation Committee - Subjective Knee Evaluation Form | 6months post procedure
Satisfaction Level | 6months post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Ivan Medina-Porqueres, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No